CLINICAL TRIAL: NCT02648958
Title: Effect of Dexmedetomidine on Ischemia-Reperfusion Injury in Unilateral Total Knee Replacement - a Randomized, Controlled Trial
Brief Title: Effect of Dexmedetomidine on Ischemia-Reperfusion Injury in Lower Extremity Operations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2015-0794
Record Dates: First submitted 2015-12-06; First posted 2016-01-07 (Estimated); Last update posted 2018-06-13 (Actual); Status verified 2016-01

CONDITIONS: Arthroplasty, Replacement
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Placebo Comparator): The control group received saline instead of dexmedetomidine.
  Interventions: Drug: normal saline
- Dexmedetomidine group (Experimental): The dexmedetomidine group received the dexmedetomidine.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The dexmedetomidine group received the dexmedetomidine infusion at a rate of 0.4mg/kg/h after a loading dose of 0.5mg/kg for 10 minutes.
  Other Names: precedex
  Arms: Dexmedetomidine group
Drug: normal saline — The control group received the normal saline infusion
  Arms: Control group

SUMMARY:
Ischemia reperfusion injury causes the release of free oxygen radicals. The selective alpha2-receptor agonist, dexmedetomidine, has an inhibitory effect on inflammatory responses during ischemic injury. The aim of this study is to evaluate the effect of dexmedetomidine on inflammatory responses during ischemia-reperfusion injury in skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesiologists classification I-III

Exclusion Criteria:

* use of antioxidants clinically significant cardiovascular, renal, or hepatic diseases heart block greater than the first degree

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
changes of malondialdehyde (μmol/L) | up to 1 day

SECONDARY OUTCOMES:
changes of interleukin-6 (pg/ml) | up to 1 day

CONTACTS AND LOCATIONS:
Overall Officials: YONGSEON CHOI, Principal Investigator — Assistant professor
Locations (1):
- Severance hospital, Seoul, South Korea